CLINICAL TRIAL: NCT00940186
Title: Clinical Pharmacokinetics Study on Pikamilone
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: center for drug metabolism and pharmacokinetics, shanghai institute of materia medica
Other Study IDs: SIMM-DMPK-080901
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- pikamilone
- dosage: low dosage group: administrate pikamilone tablet 50 mg; middle dosage group: administrate pikamilone tablet 100 mg; hige dosage group: administrate pikamilone tablet 200 mg.
- tablet

SUMMARY:
Study on the phamacokinetics of Pikamilone in healthy Chinese subject and provide informations for further phase II study.

ELIGIBILITY:
Inclusion Criteria:

* nonsmokers and in good health
* weight: BMI: 19-24
* written informed consent was finished.

Exclusion Criteria:

* disease
* taking any drug, alcohol, foods containing caffeine, or grapefruits and juice before study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 15 male subjects and 15 female subjects were enrolled in this study. They were divided into three groups by random and each group contained 5 male and 5 female subjects.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-03; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D F Zhong, PH.D, Study Chair — Shanghai Institute of Materia Medica, Chinese Academy of Sciences
Locations (1):
- the second hospital to liaoning university of TCM, Shenyang, Liaoning, China